CLINICAL TRIAL: NCT04083950
Title: Induction of Gut Permeability by an Oral Vaccine
Status: Active, not recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: USDA, Western Human Nutrition Research Center (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: FL109
Record Dates: First submitted 2019-09-05; First posted 2019-09-10 (Actual); Last update posted 2025-11-24 (Actual); Status verified 2025-11

CONDITIONS: Intestinal Permeability; Inflammation; Vaccine; Typhoid Fever
Keywords: Gastrointestinal Health; Intestinal Permeability; Inflammation; Vaccine Response; Ty21a Typhoid Vaccine; Typhoid Fever
MeSH Terms: conditions — Inflammation; Typhoid Fever | interventions — Aspirin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Single group (Experimental): All participants will receive the vaccine and aspirin.
  Interventions: Biological: Vivotif Typhoid Oral Vaccine; Drug: Aspirin (Positive Control)

INTERVENTIONS:
Biological: Vivotif Typhoid Oral Vaccine — One capsule is swallowed on alternate days, e.g. days 15, 17, 19, and 21, for a total of 4 capsules.
  Other Names: Ty21a Typhoid Oral Vaccine
Drug: Aspirin (Positive Control) — Three tablets (325 mg aspirin in each tablet or 975 mg total) are swallowed on days 2 and 3.
  Other Names: Aspirin Challenge

SUMMARY:
This study evaluates the effect of an oral typhoid vaccine on disruption of the intestinal barrier and response of the immune system. Intestinal and whole-body responses will be measured in all participants before and after the vaccine.

DETAILED DESCRIPTION:
The licensed Ty21a vaccine strain of S. enterica Typhi is routinely used by travelers to countries where typhoid is common. It is not known whether the vaccine causes measurable changes in intestinal permeability and whether changes in permeability are correlated with the magnitude of the vaccine response. In the current study, gut permeability will be measured in participants at baseline and after an aspirin challenge, which is known to disrupt intestinal permeability, and after the first, second, and fourth doses of a the Ty21a vaccine. Intestinal permeability will be measured using a three-sugar absorption test composed of lactulose, mannitol, and sucralose and by several plasma markers. Vaccine response will be measured by quantitating T cells and newly developed IgG-or IgA-secreting plasma cells specific for Ty21a.

ELIGIBILITY:
Inclusion Criteria:

* Body Mass Index (BMI) 18.5 - 29.9 kg/m2

Exclusion Criteria:

* Has HIV/AIDS or another disease that affects the immune system
* Has any kind of cancer
* Decline to take an HIV blood test
* Blood pressure greater than or equal to 140/90 mmhg
* Pregnant or lactating women
* Refusal to take a pregnancy test prior to the study
* Refusal to use a method of birth control during the study
* Allergy to vaccine components, i.e. Thimerosal and enteric-coated capsules
* Allergy to oral typhoid vaccine
* Allergy to aspirin
* Daily use of blood thinners
* Use of anti-inflammatory medications, i.e. nonsteroidal anti-inflammatory drugs (NSAID), aspirin, 3 or more times per month
* Use of sulfonamides or antibiotics in the past 30 days
* Use of anti-hypertensive drugs, i.e. beta blockers, diuretics, calcium channel blockers
* Use of anti-malaria drugs, i.e. Mefloquine, chloroquine, and proguanil
* Use of drugs that affect the immune system, i.e. immunosuppressants, immune-modifying drugs, corticosteroids, i.e. cortisone, prednisone, methylprednisolone, for 2 weeks or longer
* Is taking cancer treatment with radiation or drugs
* Greater than ten years residence in a typhoid-endemic area
* Receipt of typhoid vaccine in the last 5 years
* Receipt of any vaccine two weeks prior to receipt of Ty21a vaccine
* Individuals at increased risk of developing complications from a live, bacterial vaccine
* History of typhoid fever
* History of primary immune deficiency or autoimmune disease
* History of acute or chronic gastrointestinal (GI) disorder, i.e. Crohn's disease, irritable bowel syndrome, gastric ulcer
* Diarrheal illness (defined as passing 3 or more abnormally loose or watery stool in a 24 hour period) or persistent vomiting 2 weeks prior to the study
* History of bleeding disorder, including bleeding from the GI tract
* History of chronic illnesses, i.e. diabetes, cardiovascular disease, cancer, gastrointestinal malabsorption or inflammatory diseases, kidney disease, autoimmune disorders, HIV, liver disease, including hepatitis B and C.
* Asthma if taking medication on a daily basis
* Recent surgery (within 3 months)
* History of GI surgery
* Recent hospitalization (within 3 months)
* Acute febrile illness (within 2 weeks)
* Unwillingness to discontinue consumption of artificial sweeteners in foods or drinks, i.e. sport drinks, coconut water, "diet" drinks and foods (possibly containing sucralose)
* Not having at least one arm vein suitable for blood drawing
* Unwilling or uncomfortable with blood draws seven times in 29 days
* Regular blood or blood product donation and refusal to suspend donation
* Current participation in another research study
* Unable to fast for 12-16 hours

Ages: 18 Years to 49 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 10 (Actual)
Dates: Start 2019-12-04 (Actual); Primary Completion 2022-01-31 (Actual); Study Completion 2026-09-30 (Estimated)

PRIMARY OUTCOMES:
Change in intestinal permeability | Day 1, 3, 16, 18, and 22
  Measurement of sugar (lactulose, D-mannitol, and sucralose) excretion in urine.

SECONDARY OUTCOMES:
Antibody response to typhoid vaccination | Day 1, 18, 22, 24, and 29
  Measurement of Typhi-specific immunoglobulin G (IgG) and immunoglobulin A (IgA) plasma cells in peripheral blood using the antibody in lymphocyte supernatant assay.
T-cell response to typhoid vaccination | Day 1, 22, and 29
  Measurement of vaccine-specific cluster of differentiation 4 (CD4) and cluster of differentiation 8 (CD8) T-cells in peripheral blood mononuclear cells.
Change in markers of inflammation | Day 1, 3, 16, 18, 22, and 24
  Measurement of plasma cytokines, chemokines, and acute phase proteins by a multiplex immunoassay.
Change in intestinal fatty acid binding protein (iFABP) | Day 1, 3, 16, 18, and 22
  Measurement of plasma iFABP.
Change in D-lactate | Day 1, 3, 16, 18, and 22
  Measurement of plasma D-lactate.
Change in diamine oxidase | Day 1, 3, 16, 18, and 22
  Measurement of plasma diamine oxidase.
Change in lipopolysaccharide binding protein (LBP) | Day 1, 3, 16, 18, and 22
  Measurement of plasma LBP.
Change in citrulline | Day 1, 3, 16, 18, and 22
  Measurement of plasma citrulline.

CONTACTS AND LOCATIONS:
Overall Officials: Danielle Lemay, PhD, Principal Investigator — USDA, ARS, Western Human Nutrition Research Center
Locations (1):
- USDA, ARS, Western Human Nutrition Research Center, Davis, California, United States

IPD SHARING:
Plan to Share IPD: No